CLINICAL TRIAL: NCT06665503
Title: The Impact of Zinc and Probiotics in Preventing Pediatric Antibiotic-Associated Diarrhea in Southern Iran
Acronym: AAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Bagher Rahmati, Hormozgan University of Medical Sciences, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IR.HUMS.REC.1399.579; Hormozgan University (Other: Hormozgan University)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Antibiotic-associated Diarrhea; Diarrhea
Keywords: antibiotic-associated diarrhea; children zinc, probiotics; zinc; probiotics
MeSH Terms: conditions — Diarrhea | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomly assigned to three groups of equal size, exclusively receiving the standard antibiotic regimen or the zinc and probiotics groups
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 65 children in cotrol group (No Intervention): Only standard medication.
- 65 children in Zinc group (Experimental): The zinc group received oral zinc supplementation; 2.5 ml every 12 hours for children aged <1 year and 5 ml every 12 hours for older children.
  Interventions: Dietary Supplement: Zinc Supplement, probiotic
- 65 children in Probiotic group (Experimental): The probiotics group received oral probiotics; 1 probiotic sachet (KidiLact: Lacticaseibacillus rhamnosus, Lactobacillus reuteri, Lactobacillus acidophilus, Bifidobacterium infantis, Lactobacillus acidophilus, Bifidobacterium bifidum and Streptococcus thermophilus)
  Interventions: Dietary Supplement: Zinc Supplement, probiotic

INTERVENTIONS:
Dietary Supplement: Zinc Supplement, probiotic — received oral zinc supplementation; 2.5 ml every 12 hours for children aged <1 year and 5 ml every 12 hours for older children; the probiotics group received oral probiotics; 1 probiotic sachet
  Arms: 65 children in Probiotic group; 65 children in Zinc group

SUMMARY:
The Impact of Zinc and Probiotics in Preventing Pediatric Antibiotic-Associated Diarrhea in Southern Iran

DETAILED DESCRIPTION:
The participants will be children aged 3 months to 3 years.The zinc group received oral zinc supplementation; 2.5 ml every 12 hours for children aged <1 year and 5 ml every 12 hours for older children; the probiotics group received oral probiotics; 1 probiotic sachet; and the control group received nothing.

ELIGIBILITY:
Inclusion Criteria:

1. children aged 3 months to 3 years
2. prescribed antibiotics for various medical conditions

Exclusion Criteria:

1. Diarrhea, Dysentery
2. Underlying chronic disease

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of Antibiotic-Associated Diarrhea | 6 month
  Passing loose, watery stools three or more times a day after taking antibiotic by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: MohammadBagher Rahmati, Pediatrician, Study Director — Hormozgan University of Medical Sciences
Locations (1):
- Hormozgan University of Medical Sciences, Bandar Abbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: October 2024-January 2026
Access Criteria: For independent reviewers.